CLINICAL TRIAL: NCT03069404
Title: INSTrUCT-SCI: INdependent Observational STUdy of Cell Transplantation in SCI, an Investigator Initiated Trial
Brief Title: INSTrUCT-SCI: INdependent Observational STUdy of Cell Transplantation in SCI
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Foundation Wings For Life (Other)
Responsible Party: Sponsor
Other Study IDs: INSTrUCT-SCI
Record Dates: First submitted 2017-02-09; First posted 2017-03-03 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigation is a multi-year observational study following the completion of the open-label, single dose Phase I/II study involving transplantation of allogeneic HuCNS-SC cells into 12 subjects with thoracic spinal cord injury.

Subjects will be monitored at routine intervals for safety and preliminary efficacy for 5 years post-transplantation of the Phase I/II investigation CL-N02-SC.

ELIGIBILITY:
Inclusion Criteria:

* Must have undergone HuCNS-SC transplantation as a subject in the Phase I/II trial
* Must be able to provide written informed consent prior to any study related procedures
* Must agree to comply in good faith with all conditions of the study and to attend all required study visits
* Female subjects who are pregnant remain eligible for enrollment, but the MRI examination will not be performed during the pregnancy. Female subjects of child-bearing potential must have a negative urine pregnancy test prior to the MRI examination

Exclusion Criteria:

* Subjects have received or are receiving off-protocol immunosuppressive medications
* Subjects who after completion of CL-N02-SC have entered, or are about to enter any other interventional study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Spinal cord injured patients T2-T11
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
American Spinal Injury Association (ASIA) Impairment Scale Improvement | 36 months after transplantation of HuCNS-SC®
  Evidence of improvement in ASIA impairment scale as confirmed by neurological examination

CONTACTS AND LOCATIONS:
Overall Officials: Armin Curt, MD, Principal Investigator — Universitätsklinik Balgrist
Locations (1):
- Universitätsklinik Balgrist, Zurich, Switzerland